CLINICAL TRIAL: NCT01033149
Title: N-acetylcysteine in the Treatment of Bulimia Nervosa
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19223, 09-09-18-01; NAC in Bulimia Nervosa
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Bulimia Nervosa
MeSH Terms: conditions — Bulimia Nervosa | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- N-acetylcysteine (Other): open label N-acetylcysteine, flexible dose
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine, flexible dose 1200-2400mg/day

SUMMARY:
The specific aim of this study is to evaluate the efficacy, tolerability, and safety of N-acetylcysteine (NAC) in the treatment on bulimia nervosa.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, between the ages of 18 and 65. The patient population is expected to be predominantly made up of women based on previous research.
2. Patients will meet DSM-IV-TR criteria for BN for at least the last 6 months. These criteria are as follows:

   A. Recurrent episodes of binge eating. An episode of binge eating is characterized by both of the following:
   1. Eating, in a fixed period of time, an amount of food that is definitely larger than most people would eat under similar circumstances.
   2. A sense of lack of control over eating during the episode B. Recurrent inappropriate compensatory behavior to prevent weight gain, such as: self-induced vomiting; misuse of laxatives; diuretics; or other medications; fasting; excessive exercise.

   C. Binge-purge episodes occur at least two times a week in the last 3 months D. Self- evaluation in unduly influenced by body shape and weight E. The disturbance does not occur exclusively during episodes of anorexia nervosa.
3. Capacity to consent to the study and comply with study procedures.

Exclusion Criteria:

Criteria for exclusion from this study will be any of the following:

1. Have current body mass index (BMI) < 20kg/m2.
2. Women who are pregnant or lactating and women of childbearing potential who are not taking adequate contraceptive measures.
3. Subjects who are displaying clinically significant suicidality or homicidality.
4. A current or recent (within 6 months of the start of NAC) DSM-IV-TR diagnosis of substance abuse or dependence.
5. History of a personality disorder (eg, schizotypal, borderline, or antisocial) which might interfere with assessment or compliance with study procedures
6. Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease which could interfere with diagnosis, assessment, or treatment of BN. Patients should be biochemically euthyroid prior to entering the study.
7. DSM-IV-TR Anorexia nervosa
8. Serum potassium of ≤ 0.3mmol/L
9. Myocardial infarction within six months
10. Subjects taking more than 200 /µg of selenium per day, or 500 IU of Vitamin E /day
11. Subjects with known or suspected clinically relevant systemic medical disorder, including asthma, bronchospasm, or respiratory insufficiency.
12. Subjects who had recently used medications (<14 days) felt to be hazardous if taken with NAC (e.g. carbamazepine, nitroglycerin).
13. Subjects previously enrolled in this study; subjects who have previously been treated with NAC; subjects who have received an experimental drug or have used an experimental device within 30 days.

Subjects who are taking psychotropic medications will be allowed into the study as long as the dose of medication had been stable for 3 months before study inclusion and there are no plans to modify the dose during the study duration. Similarly, subjects evolved in psychotherapy for BN will be allowed to participate if attendance had been ongoing for at least 3 months before study entry. Subjects who changed doses of medication or started new therapy will be discontinued from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the weekly frequency of binge-purge episodes. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

REFERENCES:
- [Result] Guerdjikova AI, Blom TJ, Mori N, McElroy SL. N-acetylcysteine in bulimia nervosa--open-label trial. Eat Behav. 2013 Jan;14(1):87-9. doi: 10.1016/j.eatbeh.2012.11.001. Epub 2012 Nov 19. PMID 23265409